CLINICAL TRIAL: NCT03590431
Title: Bioavailability of Iodine in Cow's Milk in Swiss Adults
Acronym: BICOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Herter-Aeberli (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Principal Investigator, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BICOM 2018-00130
Record Dates: First submitted 2018-05-30; First posted 2018-07-18 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-01

CONDITIONS: Iodine Bioavailability
Keywords: iodine; bioavailability; milk
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Participant
Masking Description: Two of the three test drinks will consist of milk delivering extrinsic iodine or intrinsic iodine and will appear the same. These two milks will be labelled with "A" and "B" and masking will be applied to the participant only (single-blinded). The code will be held by the Study coordinator. However, for the water iodine-solution, blinding will not be possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bioavailability iodine milk (extrinsic) (Other): 300 ml whole cow's milk delivering ≈ 200 µg iodine (extrinsic iodine in milk, low protein-bound fraction)
  Interventions: Dietary Supplement: extrinsic iodine in milk
- bioavailability iodine milk (intrinsic) (Other): 300 ml whole cow's milk delivering ≈ 200 µg iodine (intrinsic iodine in milk, high protein-bound fraction)
  Interventions: Dietary Supplement: intrinsic iodine in milk
- bioavailability water iodine solution (Other): 300 ml water iodine solution delivering ≈ 200 µg iodine (water iodine solution)
  Interventions: Dietary Supplement: water iodine solution

INTERVENTIONS:
Dietary Supplement: extrinsic iodine in milk — 300 ml whole cow's milk delivering ≈ 200 µg iodine (extrinsic iodine, low protein-bound fraction) The whole cow's milk will be produced in an experimental barn feeding supplementary iodine to reach a final iodine concentration of ≈ 50 µg/L. The iodine content of the extrinsically labelled milk will be adjusted to the required concentration (same as intrinsic iodine milk) by adding iodine in form of potassium iodide.
  Arms: bioavailability iodine milk (extrinsic)
Dietary Supplement: intrinsic iodine in milk — 300 ml whole cow's milk delivering ≈ 200 µg iodine (intrinsic iodine, high protein-bound fraction) The whole cow's milk will be produced in an experimental barn feeding supplementary iodine to reach a final iodine concentration of ≈ 600 µg/L. This concentration will define final supplemental iodine given to the participants (adapting the total portion size).
  Arms: bioavailability iodine milk (intrinsic)
Dietary Supplement: water iodine solution — 300 ml water delivering ≈ 200 µg iodine (control)
  Arms: bioavailability water iodine solution

SUMMARY:
Iodine deficiency remains a global problem impairing health and development in affected populations. Although there has been remarkable global progress against iodine deficiency, mild and moderate iodine deficiency remain common globally, including European countries. Besides salt, milk and dairy products are important iodine sources in many industrialized countries, with varying contributions depending on the milk iodine concentration and the amount of milk and dairy consumed.

Iodine absorption in humans depends on the iodine species and possibly on the iodine status of the person. Very little data is available on iodine absorption or bioavailability from different dietary sources including milk. Inorganic iodide is thought to be absorbed almost completely (>90%). In contrast, only about two-thirds of some forms of organically-bound iodine are absorbed. The absorption of iodine from milk has not been quantified in humans. In this balance study, the investigators want to quantify the absorption of iodine in cow's milk in male and female adults and compare with the bioavailability from an iodine water solution (potassium iodide). The results of this study will inform on the bioavailability rate of iodine from cow's milk. Knowing the actual iodine bioavailability from milk is critical because milk and dairy products are major iodine sources in many industrialized countries.

The primary objective of this randomized, cross-over design study is to assess iodine bioavailability (measured using excretion in urine) from whole cow's milk delivering an iodine level of about 600 µg/L and compare them with a control iodine solution. The investigators will test three drinks within one subject: 1) a milk with an intrinsic iodine concentration of about 600 µg/L; 2) a milk with a naturally low iodine concentration and an added amount of potassium iodide (extrinsic iodine in milk matrix) to reach a level of about 600 µg/L (adapted to the intrinsic concentration in 1)); and 3) control iodine solution (extrinsic iodine in water matrix) with the same iodine concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 45 years
2. BMI 19-25 kg/m2
3. Current use of iodized salt at home
4. Signed informed consent

Exclusion Criteria:

1. Inadequate iodine status (defined as UIC <70 µg/L or >300 µg/L and assessed during screening from 5 urine spot samples)
2. Exposure to iodine-containing X-ray/ computed tomography contrast agent
3. Use of iodine-containing disinfectants (betadine)
4. History of thyroid disease (according to the participants own statement)
5. Any metabolic, gastrointestinal or chronic disease such as diabetes, hepatitis, hypertension, or cancer (according to the participants own statement)
6. Chronic use of medications (except for contraceptives)
7. Use of iodine containing supplements within 1 month prior to study start
8. Pregnancy (according to the participants own statement but confirmed by a pregnancy test with the first urine spot sample from screening)
9. Breast feeding
10. Vegan diet
11. Drug abuse
12. Extensive alcohol intake, defined as more than 3 (men) or 2 (women) standard drinks per day (i.e. 3dl beer, 1dl wine, 3-4cl liquor), with less than 2 days per week without alcohol consumption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Iodine concentration in urine | Days 1, 2, 3, 8, 9, 10, 15, 16 and 17
  measured by Sandell-Kolthoff method, mikrograms per liter To calculate iodine absorption, excretion and retention.

SECONDARY OUTCOMES:
TSH | day 1
  thyroid function test at baseline
T4 | day 1
  thyroid function test at baseline
iodine content of standardized diet | prior to study start
  the quantitative assessment of iodine content in the participants' standardized diet

OTHER OUTCOMES:
Age | at screening
  Age in years
BMI | at screening
  BMI calculated from measured weight and height

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, Dr., Principal Investigator — University of Zurich
Locations (1):
- ETH Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Reijden OL, Galetti V, Burki S, Zeder C, Krzystek A, Haldimann M, Berard J, Zimmermann MB, Herter-Aeberli I. Iodine bioavailability from cow milk: a randomized, crossover balance study in healthy iodine-replete adults. Am J Clin Nutr. 2019 Jul 1;110(1):102-110. doi: 10.1093/ajcn/nqz092. PMID 31788697